CLINICAL TRIAL: NCT01490658
Title: A Randomized, Single-Blind, Three-Period Crossover Study Examining the Single Dose Pharmacokinetics of Concomitantly Administered Repaglinide and Metformin Versus Combination Tablet Dosing (NN4440) in Fed Healthy Volunteers
Brief Title: Single Dose Pharmacokinetics of Repaglinide, Metformin and Combination Tablet in Fed Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NN4440-1753
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment period 1 (Experimental)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet
- Treatment period 2 (Experimental)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet
- Treatment period 3 (Active Comparator)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet

INTERVENTIONS:
Drug: repaglinide — Single dose of 2 mg tablets administered immediately prior to a standard high fat breakfast concomitantly with metformin as separate tablets. Subjects will be randomised to receive trial drug on 3 separate dosing visits in varying order out of 6 possible treatment periods
Drug: metformin — Single dose of 500 mg tablets administered immediately prior to a standard high fat breakfast concomitantly with repaglinide as separate tablets. Subjects will be randomised to receive trial drug on 3 separate dosing visits in varying order out of 6 possible treatment periods
Drug: repaglinide and metformin combination tablet — Single dose of 2 mg repaglinide/500 mg metformin (NN4440 2/500) or 1 mg repaglinide/500 mg metformin (NN4440 1/500)administered immediately prior to a standard high fat breakfast. Subjects will be randomised to receive trial drug on 3 separate dosing visits in varying order out of 6 possible treatment periods

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare repaglinide and metformin as co-administered tablets and as a combination tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers (female not pregnant, lactating or breastfeeding)
* BMI (Body Mass Index) between 19-29 kg/m^2, both inclusive
* Fasting plasma glucose from 70-115 mg/dl
* Subject is judged to be in good health on the basis of their medical history, physical examination, ECG (electrocardiogram), and routine laboratory data

Exclusion Criteria:

* Any clinically significant disease history, in the opinion of the Investigator, of systemic or organ disease
* Clinically significant abnormalities on pre-study clinical examination or any laboratory measurements during screening
* Positive results on screening for Hepatitis B surface antigen, Hepatitis C antibody and HIV (human immunodeficiency virus) antibody
* Positive results on the drug abuse/alcohol screen
* Any regular use of prescription or nonprescription drugs, including mega-vitamin or herbal supplement regimens, other than contraceptives, that cannot be stopped at least 1 week prior to Visit 2 (trial product dose administration) and for the duration of the study
* Subject is currently a smoker (more than one cigarette per day or equivalent)
* Use of grapefruit or grapefruit juice within 7 days of trial product dose administration
* Blood donation, surgery or trauma with significant blood loss (500 mL) within the last 2 months prior to dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Repaglinide and metformin AUC (Area under the Curve) fed state concomitant tablet administration
Repaglinide and metformin AUC (Area under the Curve) NN4440 (2/500) combination tablet
Repaglinide and metformin Cmax (maximum plasma concentration) fed state concomitant tablet administration
NN4440 (2/500) Cmax (maximum plasma concentration) combination tablet

SECONDARY OUTCOMES:
Repaglinide AUC after NN4440 (1/500) during fed state
Repaglinide Cmax after NN4440 ((1/500) during fed state
Change in physical examinations from screening
Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Austin, Texas, United States

REFERENCES:
- [Result] Hoelscher D, Chu PL, Lyness W. Fixed-dose combination tablet of repaglinide and metformin is bioequivalent to concomitantly administered individual tablets of repaglinide and metformin : randomized, single-blind, three-period crossover study in healthy subjects. Clin Drug Investig. 2008;28(9):573-82. doi: 10.2165/00044011-200828090-00004. PMID 18666804
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com